CLINICAL TRIAL: NCT02945969
Title: Effect of Dietary Sodium Reduction in Kidney Disease Patients With Albuminuria
Brief Title: Sodium Lowering and Urinary Protein Reduction Trial
Acronym: SUPER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tulane University School of Public Health and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Katherine T Mills, Assistant Professor, Tulane University School of Public Health and Tropical Medicine
Organization: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1P20GM109036-P1; 1P20GM109036 (NIH)
Record Dates: First submitted 2016-10-25; First posted 2016-10-26 (Estimated); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Chronic Kidney Disease; Albuminuria
Keywords: dietary sodium; albuminuria; chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Albuminuria | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Sodium Diet (Experimental): Behavioral modification to decrease dietary sodium intake to ≤2,300 mg/day for 24 weeks. The intervention program consists of two phases. An initial 12-week intensive phase will include weekly individual and group sessions. This will be followed by a 12-week maintenance phase that includes telephone counseling sessions every 2 weeks.
  Interventions: Behavioral: Low Sodium Diet
- Usual Diet (No Intervention): No dietary intervention.

INTERVENTIONS:
Behavioral: Low Sodium Diet — Once randomized to the Intervention program, study participants will be grouped into intervention cohorts of approximately 10 participants per group to facilitate group counseling sessions. Both the intensive intervention phase and the maintenance phase will include individual and group behavioral modification counseling designed to facilitate a reduction in dietary sodium intake. Success of the intervention will be assessed by comparing the urine sodium measurements from 24-hour urine collections performed at screening, 12 weeks and 24 weeks.
  Arms: Low Sodium Diet

SUMMARY:
The proposed randomized controlled trial will test the effect of dietary sodium reduction on albuminuria in patients with proteinuric chronic kidney disease. Results from this study will clarify the role of dietary sodium reduction in management of patients with proteinuric chronic kidney disease and its potential to halt the progression of chronic kidney disease.

DETAILED DESCRIPTION:
Proteinuria is an early and sensitive marker of kidney damage and a risk factor for chronic kidney disease (CKD) progression, cardiovascular disease and all-cause mortality. Several cross-sectional epidemiological studies have reported an association between sodium intake and albuminuria (majority of proteinuria) that is independent of blood pressure (BP). In addition, a handful of small clinical trials have suggested a reduction in dietary sodium intake may decrease albuminuria in patients with CKD. The overall goal of this randomized controlled trial is to study the effect of dietary sodium reduction on albuminuria in CKD patients with albuminuria. A total of 150 participants with CKD and albuminuria will be recruited and randomly assigned to either a 24-week intensive behavioral modification program designed to reduce dietary sodium intake to 2,300 mg/day or to usual care in a 1:1 randomization ratio. The primary outcome will be the difference between the active intervention and control groups for change in urinary albumin-to-creatinine ratio from baseline to 24 weeks of follow-up. Urinary albumin-to-creatinine ratio will be assessed as the average of two 24-hour urine collections at each time point. Secondary outcomes will include estimated glomerular filtration rate (eGFR), BP, and number of antihypertensive medications. Urinary sodium excretion will be used to measure the success of the intervention. Racial differences in albuminuria changes due to reduction in dietary sodium intake will be analyzed. The intervention program will be modeled on best practices derived from the investigators prior experience in conducting sodium reduction behavioral interventions. The intervention program will address individual barriers to long-term sodium reduction and generate collective enthusiasm and motivation for adherence to the program. Study staff will receive training and direct support from a consultant with extensive experience in successful implementation of behavioral and dietary modification interventions. Results from this study will clarify the role of dietary sodium reduction in management of CKD patients with albuminuria and its potential to halt the progression of CKD, a global public health concern. The study will also explore the interaction of race/ethnicity with dietary sodium reduction on albuminuria in CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 21 years of age: The lower age limit was chosen based on the National Institutes of Health (NIH) definition of adults for participation in research
* Any race or ethnicity: The investigators expect to recruit 50-60% African American and 40-50% non-African American (White, Hispanic, and Asian Americans), with the vast majority of the latter being non-Hispanic Whites.
* eGFR < 90 mL/min/1.73m2 but > 30 mL/min/1.73m2. The upper limit for eGFR was chosen to include participants with a clinically significant decrease in renal function. The investigators chose an upper eGFR limit slightly higher than the Kidney Disease Outcomes Quality Initiative (KDOQI) definition of moderately reduced glomerular filtration rate (GFR) to be more inclusive of patients with mild reduction in GFR but significant proteinuria. The lower eGFR limit was set to exclude patients with advanced CKD, where the potential effects of dietary sodium reduction on proteinuria may not be apparent or greatly alter CKD progression. The eGFR to define eligibility will be calculated using calibrated serum creatinine values and the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) estimating equation.
* Albumin-to-creatinine ratio > 30mg/g

Exclusion Criteria:

* Albuminuria ≥1.5 g/g or kidney structural change
* Prior kidney transplant based on self-report
* Immunosuppression or other immunotherapy within the past six months prior to enrollment based on patient self-report
* History of cancer other than non-melanoma skin cancer within two years prior to enrollment based on patient self-report
* History of polycystic kidney disease
* Currently receiving dialysis treatment
* History of human immunodeficiency virus (HIV)
* Current pregnancy, breastfeeding or plans to become pregnant during the study
* Consumption of ≥14 alcoholic drinks/week or consumption of ≥6 drinks/occasion
* Current participation in another lifestyle intervention trial
* Current residence or planned residence make it difficult to meet trial requirements
* Other concerns regarding ability to meet trial requirements, at the discretion of the principal investigator

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2016-11; Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Net Change in Urinary Albumin-to-Creatinine Ratio (ACR) | Assessed twice at baseline, once at week 12, and twice at week 24

SECONDARY OUTCOMES:
Net Change in Urinary Albumin | Assessed twice at baseline, once at week 12, and twice at week 24
Estimated Glomerular Filtration Rate (eGFR) | Assessed at baseline, week 12, and week 24
Blood Pressure | Assessed twice at baseline, once at week 12, and twice at week 24
Number of Antihypertensive Medications | Assessed at baseline, week 12, and week 24

CONTACTS AND LOCATIONS:
Overall Officials: Katherine T Mills, PhD, MSPH, Principal Investigator — Tulane University School of Public Health and Tropical Medicine
Locations (1):
- Tulane University, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McMahon EJ, Campbell KL, Bauer JD, Mudge DW, Kelly JT. Altered dietary salt intake for people with chronic kidney disease. Cochrane Database Syst Rev. 2021 Jun 24;6(6):CD010070. doi: 10.1002/14651858.CD010070.pub3. PMID 34164803